CLINICAL TRIAL: NCT02916693
Title: Mirabegron For Erectile Dysfunction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00097439
Record Dates: First submitted 2016-09-22; First posted 2016-09-27 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Erectile Dysfunction; Overactive Bladder; Urinary Incontinence
Keywords: Mirabegron; Overactive Bladder; Erectile Dysfunction; Beta 3 agonist
MeSH Terms: conditions — Erectile Dysfunction; Urinary Bladder, Overactive; Urinary Incontinence | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mirabegron (Experimental): Participants take 25- 50mg oral Mirabegron tablets daily for 12 weeks,
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — FDA-approved, beta 3 agonist for over active bladder
  Other Names: Myrbetriq

SUMMARY:
The only class of oral erectile dysfunction (ED) medication on the market are the phosphodiesterase Type 5 inhibitors (PDE5i). This pilot study is being done to evaluate the effect of Mirabegron, an oral beta-3 adrenergic agonist, on men with both Overactive Bladder (OAB) symptoms and mild to moderate ED.

DETAILED DESCRIPTION:
ED affects up to 30 million men in the United States. The only class of oral medication approved for ED is PDE5i. These include sildenafil, tadalafil, vardenafil and avanafil. Other pharmacologic options in the treatment of ED are delivered as an intraurethral suppository (alprostadil) or intracavernosal injection (alprostadil, papaverine, phentolamine, atropine). These are more invasive routes of administration. Men who fail to obtain benefit from a PDE5i or those who have a contraindication to this class of medication may ultimately avoid further pharmacologic treatment options. An alternative class of oral medication to treat ED may prove to be of benefit to a large population of underserved men.

There is in vitro evidence that beta-3 adrenergic receptors exist in human corpus cavernosum tissue. Activation of these receptors results in vasorelaxation, suggesting a potential pro-erectogenic effect is possible in vivo. Additionally, nebivolol, a beta-blocker, has pro-erectogenic effects noted in several studies. There is evidence that nebivolol exerts beta-3 adrenergic agonism, which may explain the mechanism by which these effects occur.

Mirabegron is the only available beta-3 adrenergic agonist in the United States. Its favorable safety profile and the potential for therapeutic efficacy in ED make it suitable for further investigation.

It is hypothesized that beta-3 adrenergic activation offers a pharmacologic target for the treatment of ED. Men with mild, mild to moderate, or moderate ED and symptoms of OAB can be recruited with pre- and post- Mirabegron administration assessment of their ED to determine the validity of this hypothesis. Men with severe ED will be excluded as historical data shows they are less likely to benefit from oral pharmacologic therapy alone. Mirabegron is approved by the U.S. Food and Drug Administration (FDA) for the treatment of adults with OAB.

ELIGIBILITY:
Inclusion Criteria:

* presence of mild ED [Erectile Function domain of the International Index of Erectile Function (IIEF EF) score 22-25], mild to moderate ED (IIEF EF domain score 17-21) or moderate ED (IIEF EF domain score 11-16)
* presence of OAB symptoms for at least 3 months
* at least 3 micturitions per day
* at least 3 episodes of urgency in a 3 day period

Exclusion Criteria:

* history of pelvic surgery
* concurrent ED therapy
* history of penile surgery
* history of priapism (unwanted, prolonged painful erection)
* history of neurologic disease
* uncontrolled hypertension: systolic blood pressure (BP) > 140 mmHg or diastolic BP > 90 mmHg
* Stage 4 or 5 chronic kidney disease, Creatinine clearance rate < 30ml/min
* moderate or severe hepatic impairment
* concomitant use of CYP2D6-metabolized drugs or digoxin
* post void residual greater than 150 ml
* evidence of urinary tract infection on urinalysis and/or urine culture

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur L Burnett, M.D., M.B.A., Principal Investigator — Johns Hopkins, School of Medicine
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirabegron 25 mg to 50 mg Treatment: Single-center, non-randomized, single-arm study
Period: Overall Study
Arm/Group | Mirabegron 25 mg to 50 mg Treatment
Started | 20
Completed | 13
Not Completed | 7
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Groups:
- Mirabegron 25 mg to 50 mg Treatment: Single-center, non-randomized, single-arm study Participants received Mirabegron 25 mg for 2 weeks and switched to the 50 mg for 10 weeks
Arm/Group | Mirabegron 25 mg to 50 mg Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (6.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Co-morbidities [Count of Participants; unit: Participants]
  Diabetes Mellitus | 2
  Hypertension | 8
  Hyperlipidemia | 8
  Cardiovascular disease | 2
Smoking History [Count of Participants; unit: Participants]
  Never Smoker | 10
  Current Smoker | 3
  Ex-smoker | 7
Erectile Dysfunction (ED) Severity [Count of Participants; unit: Participants] — ED Severity classified as mild, mild to moderate and moderate.
  Participants
    Mild | 3
    Mild to moderate | 6
    Moderate | 11

OUTCOME MEASURES:

1. Primary Outcome: Erectile Function Assessed by IIEF Questionnaire
Description: The International Index for Erectile Function (IIEF) questionnaire will be administered. This is a 15 item tool; 6 ask questions addressing Erectile function. Scores from 0-30 can be obtained in this domain. Scores are interpreted as follows: 0-6 = Severe dysfunction, 7-12 = Moderate dysfunction, 13-18 = mild-moderate dysfunction, 19-24 = mild dysfunction, 25-30 = No dysfunction.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Mirabegron: Baseline IIEF scores of participants
Arm/Group | Mirabegron
Number analyzed (Participants) | 20
score on a scale | 12.7 (5.4)

2. Primary Outcome: Erectile Function Assessed by IIEF Questionnaire
Description: as for outcome 1
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Mirabegron: Participants received Mirabegron 25 mg treatment.
Arm/Group | Mirabegron
Number analyzed (Participants) | 13
score on a scale | 13.8 (5.1)

3. Primary Outcome: Erectile Function Assessed by IIEF Questionnaire
Description: as for outcome 1
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Mirabegron: Participants received Mirabegron 50 mg treatment.
Arm/Group | Mirabegron
Number analyzed (Participants) | 13
score on a scale | 15.3 (4.2)

4. Primary Outcome: Erectile Function Assessed by IIEF Questionnaire
Description: as for outcome 1
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirabegron
Number analyzed (Participants) | 13
score on a scale | 17.8 (7.9)

5. Primary Outcome: Erectile Function Assessed by IIEF Questionnaire
Description: as for outcome 1
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirabegron
Number analyzed (Participants) | 13
score on a scale | 15.8 (6.9)

6. Secondary Outcome: Health Related Quality of Life as Assessed by the OAB Questionnaire
Description: The Overactive Bladder questionnaire (OAB-q) health-related quality of life (HRQL) form will be administered. It is a 13 item tool assessing the health-related quality of life (HRQL) impact of OAB. Scores range from 13 to 78 with higher scores indicating a greater degree of a lower quality of life due to OAB.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Mirabegron: Baseline score of OAB-q
Arm/Group | Mirabegron
Number analyzed (Participants) | 20
score on a scale | 35.3 (13.6)

7. Secondary Outcome: Health Related Quality of Life as Assessed by the OAB Questionnaire
Description: as for outcome 6
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirabegron
Number analyzed (Participants) | 13
score on a scale | 30.7 (11.4)

8. Secondary Outcome: Health Related Quality of Life as Assessed by the OAB Questionnaire
Description: as for outcome 6
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirabegron
Number analyzed (Participants) | 13
score on a scale | 30. (13.3)

9. Secondary Outcome: Health Related Quality of Life as Assessed by the OAB Questionnaire
Description: as for outcome 6
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirabegron
Number analyzed (Participants) | 13
score on a scale | 26.9 (10.6)

10. Secondary Outcome: Health Related Quality of Life as Assessed by the OAB Questionnaire
Description: as for outcome 6
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirabegron
Number analyzed (Participants) | 13
score on a scale | 27.9 (14.7)

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Mirabegron 25 mg to 50 mg: Single-center, non-randomized, single-arm study Participants received Mirabegron 25 mg for 2 weeks and switched to the 50 mg for 10 weeks.
Arm/Group | Mirabegron 25 mg to 50 mg
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 5/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mirabegron 25 mg to 50 mg (N=13)
Headache (General disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Back or leg pain (Musculoskeletal and connective tissue disorders) | 1
Flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
Among the limitations of this study are the small number of subjects, short duration of therapy, and a single-arm design with no control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-05-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT02916693/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT02916693/ICF_001.pdf